CLINICAL TRIAL: NCT03027895
Title: Endoscopic Ultrasound-guided Drainage of Walled Off Necrosis (WON)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yiqi Du (Other)
Responsible Party: Sponsor-Investigator, Yiqi Du, Professor, Changhai Hospital
Organization: Changhai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017010302
Record Dates: First submitted 2017-01-14; First posted 2017-01-23 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Pancreatic Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumen-apposing metal stent(LAMS) (Experimental): Lumen-apposing metal stent(LAMS) will be deployed by endoscopist under the guidance of EUS
  Interventions: Device: Lumen-apposing metal stent (LAMS)
- Double pigtail plastic stent(DPPS) (Active Comparator): Double pigtail plastic stent(DPPS) will be deployed by endoscopist under the guidance of EUS
  Interventions: Device: Double pigtail plastic stent (DPPS)

INTERVENTIONS:
Device: Lumen-apposing metal stent (LAMS) — Endoscopic Ultrasound-guided Drainage of WON with LAMS
  Arms: Lumen-apposing metal stent(LAMS)
Device: Double pigtail plastic stent (DPPS) — Endoscopic Ultrasound-guided Drainage of WON with DPPS
  Arms: Double pigtail plastic stent(DPPS)

SUMMARY:
The purpose of this study is to compare the effect of lumen-apposing metal stent (LAMS) and double pigtail plastic stents (DPPSs) on the drainage of pancreatic walled-off necrosis (WON), mainly to observe the efficacy and safety of LAMS for WON.

DETAILED DESCRIPTION:
Patient with pancreatic walled-off necrosis (WON) would be treated randomized with lumen-apposing metal stent (LAMS) or double pigtail plastic stents (DPPSs) under the guidance of Endoscopic Ultrasonography. The investigators compare the effect of the two stents, including technical success, clinical success, adverse event, recurrence, and so on.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with ages from 18-80 years old
2. Subject with pancreatic pseudocysts confirmed by CT
3. Subject with a history of MSAP or SAP, the pseudocysts were formed more than 3 months
4. The size of pseudocyst is more than 6 cm, and the cyst adjacent to the gastric wall
5. Subject has the symptoms related with the pseudocyst
6. The consent form has been signed

Exclusion Criteria:

1. Subject is younger than 18 years or older than 80 years
2. Pancreatic pseudocyst communicate with the main pancreatic duct
3. Subject can't accept the endoscopic procedure
4. Pancreatic pseudocyst with infection or subject diagnosed with pancreatic abscess
5. The distance between gastric and the wall of the pseudocyst is more than 1 cm
6. Subject with 2 or more than 2 cysts
7. Subject has blood coagulation dysfunction
8. Pregnant or subject has mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
clinical success | uo to 1 months
  The cysts completely disappeared, or diameter ≤ 2cm in the imaging follow-up symptoms have eased

SECONDARY OUTCOMES:
adverse event | up to 2months/ stent remove
  any adverse event occured after stent inserted
recurrence rate | up to 12 months
  After the clinical success, imaging examination show cyst again and accompanied by symptoms
technical success | up to 48 hours
  Stent placed through the wall bracket and pancreatic pseudocyst successfully

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu HY, Xie P, Song YX, Li ZS, Jin ZD, Du YQ. Lumen-apposing metal stents (LAMS) versus plastic stents for EUS-guided drainage of walled-off necrosis (WON) (LVPWON): study protocol for a multicenter randomized controlled trial. Trials. 2018 Oct 11;19(1):549. doi: 10.1186/s13063-018-2901-3. PMID 30305160